CLINICAL TRIAL: NCT03423654
Title: Spatial Cognitive Training in Visual Impairment
Brief Title: Spatial Cognitive Training
Acronym: SCTVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed out due to recruitment complications.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C2243-P
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Blind

STUDY DESIGN:
Intervention Model Description: Spatial Training group and Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group (Experimental): Spatial training
  Interventions: Other: Spatial Training
- Control Group (Other): Letter number matching
  Interventions: Other: Letter number matching

INTERVENTIONS:
Other: Spatial Training — Spatial Training using a 5x5 grid
  Arms: Training Group
Other: Letter number matching — Letter number matching
  Arms: Control Group

SUMMARY:
This study is designed to see if doing regular training on a spatial imagery task leads to improvements in the ability to do the trained spatial imagery task and in the ability to get around in everyday activities.

DETAILED DESCRIPTION:
The investigators will recruit 40 blind participants, randomized by the investigators' CVNR statistician into two groups. One group will undergo the experimental intervention (spatial cognitive training) and the other will undergo a control intervention involving letter-number matching. The participants will include women and minorities in proportion to the demographics of the Veteran population attending the Atlanta VA.

ELIGIBILITY:
Inclusion Criteria:

* Inability to perceive visual stimuli, i.e. no light perception, with stable visual loss over the past year
* The investigators anticipate that causes of blindness will be ocular, including:

  * glaucoma
  * diabetic retinopathy and macular degeneration
  * the most common causes of blindness in Veterans
  * as well as possibly late-onset Leber's optic atrophy and ocular trauma (in the absence of TBI)
* To minimize heterogeneity due to variations in age and the duration of visual loss, the investigators will restrict enrollment to Veterans and Non-Veterans over the age of 50 who lost light perception within the last 5 years, and who have completed standard O&M training.
* From a practical standpoint, this also enables the investigators to focus on participants who can potentially benefit most from the proposed intervention.

Exclusion Criteria:

* Participants will be excluded if they have any neurological condition, such as:

  * TBI
  * history of blast exposure
  * stroke
  * brain tumors
  * epilepsy, etc.
* Participants will also be excluded if MRI scanning is contra-indicated, e.g.:

  * due to an implanted device such as a pacemaker
  * or foreign bodies of ferromagnetic nature
* Cognitive screening will be performed using the Repeatable Battery for Assessment of Neuropsychological Status (RBANS, Randolph, 1998) and participants with cognitive impairment will be excluded based on a score of 1.5 SD below the mean for the Verbal Memory Index.
* The investigators will test participants' hearing using a validated screening questionnaire (Screening Version of the Hearing Handicap Inventory for the Elderly, HHIE-S, Wentry & Weinstein, 1983, Lichtenstein et al., 1988) followed by assessment of audiometric pure tone (0.5, 1.0, 2.0, 4.0 KHz) hearing thresholds in the CVNR sound booth.
* Participants with more than mild hearing loss (HHIE score >8 or audiometric thresholds >40dB) will be excluded (Wentry & Weinstein, 1983; Wilson, 2009), given that the investigators are relying on audio cues.
* The investigators will also exclude visually impaired Veterans who are dependent on a wheelchair or scooter for mobility, as they will not be able to take part in the real-world task.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: April Y. Maa, MD BS, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Training Group | Control Group
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Training Group | Control Group | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Spatial Ability
Description: Ability to orient to where participants began at the beginning of task. Using a 5x5 grid on testing device, a 5x5 grid that the participant will have to walk, and a 5x5 grid during task in MRI.
Time Frame: 1 month
Population: Study terminated early and not enough data collected to be able to run proper analysis. Some data lost due to machine malfunction. Statistics was not able to be performed due to lost data.
Arm/Group | Training Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 4 week per participant.
Arm/Group | Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03423654/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03423654/Prot_SAP_001.pdf